CLINICAL TRIAL: NCT01974258
Title: A PHASE Ib, OPEN-LABEL STUDY EVALUATING THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF ONARTUZUMAB IN COMBINATION WITH VEMURAFENIB AND/OR COBIMETINIB IN PATIENTS WITH ADVANCED SOLID MALIGNANCIES
Brief Title: Safety, Tolerability, and Pharmacokinetics of Onartuzumab Combined With Vemurafenib and/or Cobimetinib in Cancer Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29026
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — cobimetinib; onartuzumab; Vemurafenib

ARMS (4):
- Dose-expansion: onartuzumab + cobimetinib (Experimental)
  Interventions: Drug: Cobimetinib; Drug: Onartuzumab
- Dose-expansion: onartuzumab + vemurafenib (Experimental)
  Interventions: Drug: Onartuzumab; Drug: Vemurafenib
- Dose-expansion: onartuzumab + vemurafenib + cobimetinib (Experimental)
  Interventions: Drug: Cobimetinib; Drug: Onartuzumab; Drug: Vemurafenib
- Dose-finding: onartuzumab + vemurafenib + cobimetinib (Experimental)
  Interventions: Drug: Cobimetinib; Drug: Onartuzumab; Drug: Vemurafenib

INTERVENTIONS:
Drug: Cobimetinib — Escalating dose
  Arms: Dose-finding: onartuzumab + vemurafenib + cobimetinib
Drug: Cobimetinib — Orally administered once daily for 21 consecutive days, followed by 7 days off.
  Arms: Dose-expansion: onartuzumab + cobimetinib; Dose-expansion: onartuzumab + vemurafenib + cobimetinib
Drug: Onartuzumab — Administered by IV infusion every 2 weeks
Drug: Vemurafenib — Orally administered twice daily
  Arms: Dose-expansion: onartuzumab + vemurafenib; Dose-expansion: onartuzumab + vemurafenib + cobimetinib; Dose-finding: onartuzumab + vemurafenib + cobimetinib

SUMMARY:
This study will evaluate the maximum tolerated dose and dose-limiting toxicities of vemurafenib and/or cobimetinib when used with onartuzumab in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >/= 18 years of age.
* Patients with histologically confirmed, BRAFV600-mutant, unresectable, locally advanced or metastatic solid malignancies. OR
* Patients with a histologically confirmed, KRAS-mutant, Stage IV colorectal adenocarcinoma, or KRAS-mutant metastatic non-small-cell lung carcinoma. OR
* Patients with histologically confirmed BRAFV600-mutant unresectable Stage IIIC or Stage IV metastatic melanoma.
* Valid MET IHC test result.
* Measurable disease per Response Evaluation Criteria in Solid Tumors v1.1
* ECOG performance status of 0 or 1.
* For BRAFV600-mutant cancers:
* Previously untreated for their melanoma or previously treated for their melanoma but without prior exposure to any HGF, MET, BRAF, or MEK inhibitor therapy
* BRAFV600-mutant solid malignancies other than melanoma for which standard therapy does not exist has proven to be ineffective or intolerable or is considered inappropriate.

Patients must not have had prior exposure to HGF, MET, BRAF, or MEK inhibitor therapy.

* For KRAS-mutant cancers:
* mCRC patients must have received therapeutic regimens including oxaliplatin, irinotecan, 5-FU, and bevacizumab, or determined to be ineligible for these treatments. Patients must not have had prior exposure to HGF, MET, BRAF, or MEK inhibitor therapy.
* Metastatic NSCLC patients must have received platinum-based doublet chemotherapy or determined to be ineligible for this regimen. Patients must not have had prior exposure to HGF, MET, BRAF, or MEK inhibitor therapy.
* Consent to provide tumor tissue for biomarker analyses.
* Life expectancy >/= 12 weeks.
* Fully recovery from the effects of any major surgery or significant traumatic injury within 14 days from the first dose of study treatment.
* Adequate hematologic and end organ function, as defined by clinical laboratory results.
* Use of effective form(s) of contraception as defined by protocol during the course of this study and for at least 6 months after study drug discontinuation.

Exclusion Criteria:

* Palliative radiotherapy or experimental therapy within 28 days prior to first dose of study drug treatment.
* Major surgical procedure or significant traumatic injury from 28 days prior to first dose of study drug treatment until end of study.
* History of another malignancy in the previous 5 years, unless cured by surgery alone and continuously disease free. Exceptions include appropriately treated cervical carcinoma in situ, non-melanoma skin carcinoma, Stage I uterine cancer, localized prostate cancer that has been treated surgically and is presumed cured, or other malignancies with an expected curative outcome.
* Brain metastasis or spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated central nervous system (CNS) metastases or spinal cord compression without evidence of clinically stable disease for more than 14 days.

Note: Patients with treated CNS metastases who are asymptomatic and on a stable dose of corticosteroids for more than 14 days prior to Cycle 1 Day 1 are eligible.

* For patients given cobimetinib: Evidence of visible retinal pathology that is considered a risk factor for neurosensory detachment, retinal vein occlusion, or neovascular macular degeneration, or of conditions that are risk factors for retinal vein occlusion.
* Current or history of clinically significant cardiac or pulmonary dysfunction.
* Lack of recovery to Grade 1 or better from adverse events due to investigational or other agents administered more than 28 days prior to enrollment, except for alopecia.
* Current severe, uncontrolled systemic disease.
* Inability or unwillingness to swallow pills.
* History of malabsorption or other condition that would interfere with gastrointestinal absorption of study drug.
* History of clinically significant liver disease, current alcohol abuse, or known infection with HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV).
* Severe (Grade 3 and above) active infection at enrollment, or other serious underlying medical conditions.
* Required medication known to cause edema and/or cardiac failure.
* Active autoimmune disease.
* Uncontrolled ascites requiring weekly, large-volume paracentesis for 3 consecutive weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence of dose-limiting toxicities (DLTs) of vermurafenib and/or cobimetinib used in combination with onartuzumab. | 24 to 36 months
Safety: Incidence of anti-therapeutic antibodies against onartuzumab. | 24 to 36 months
Safety: Incidence of adverse events (AE) | 24 to 36 months

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum concentration (Cmax) of onartuzumab | 24 to 36 months
Pharmacokinetics: Maximum concentration (Cmax) of cobimetinib | 24 to 36 months
Pharmacokinetics: Maximum concentration (Cmax) of vemurafenib | 24 to 36 months
Efficacy: Overall response rate | 24 to 36 months
Efficacy: Progression-free survival | 24 to 36 months
Efficacy: Duration of response | 24 to 36 months
Efficacy: Overall survival | 24 to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- United States (6):
  - Los Angeles, California
  - Sarasota, Florida
  - Detroit, Michigan
  - Canton, Ohio
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee